CLINICAL TRIAL: NCT02755493
Title: Quantifying and Developing Countermeasures for the Effect of Fatigue-Related Stressors on Automation Use and Trust During Robotic Supervisory Control"
Brief Title: Quantifying and Developing Countermeasures for the Effect of Fatigue-Related Stressors on Automation Use and Trust During Robotic Supervisory Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Space Biomedical Research Institute (Other)
Responsible Party: Principal Investigator, Elizabeth B. Klerman, Associate Professor, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HFP04201
Record Dates: First submitted 2016-04-18; First posted 2016-04-29 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Sleep Deprivation
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sleep Deprivation (Experimental): Sleep deprivation
  Interventions: Behavioral: Sleep deprivation

INTERVENTIONS:
Behavioral: Sleep deprivation

SUMMARY:
This project proposes to both develop and test adaptive automation countermeasures for the effects of stressors such as sleep deprivation (SD) on human performance related to robotic tasks, and investigate the relationship between human trust and appropriate use of these countermeasures.

ELIGIBILITY:
Inclusion Criteria:

* healthy by history, physical exam, laboratory evaluations of urine and blood, electrocardiogram (ECG), psychological screening, and self-reported sleep quality.
* engineering or computer programming experience

Exclusion Criteria:

* color blind
* pregnant or nursing
* using any prescription or non-prescription medications, caffeine, alcohol or tobacco for the three weeks prior to beginning the inpatient experiments

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Performance metrics on simulated robotic tasks - time | 72 hours
  Over this 72 hour time frame there will be six assessments. Once on Day1, 4 times during the sleep deprivation on Days 2-3, and once on Day 4, the participant will perform computer simulations of "missions" with tasks. The time to complete tasks will be one of the metrics. The change in metrics related to length of time of awake will be assessed using longitudinal analysis methods.
Performance metrics on simulated robotic tasks - number complete | 72 hours
  Over this 72 hour time frame there will be six assessments Once on Day1, 4 times during the sleep deprivation on Days 2-3, and once on Day 4, the participant will perform computer simulations of "missions" with tasks. The number of completed tasks will be one of the metrics.The change in metrics related to length of time of awake will be assessed using longitudinal analysis methods.
Performance metrics on simulated robotic tasks - resources uses | 72 hours
  Over this 72 hour time frame there will be six assessments Once on Day1, 4 times during the sleep deprivation on Days 2-3, and once on Day 4, the participant will perform computer simulations of "missions" with tasks. The resources used will be one of the metrics.The change in metrics related to length of time of awake will be assessed using longitudinal analysis methods.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth B Klerman, MD PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States